CLINICAL TRIAL: NCT07366944
Title: PCOS and Problem of Eye Dryness: Is There a Benefit From Lifetyle Changes in Obese Women
Brief Title: PCOS and Problem of Eye Dryness: Is There a Benefit From Lifetyle Changes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB000-14233-63
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome; Dry Eye; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Dry Eye Syndromes; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): twenty females with PCOS, eye dryness , and obesity will receive metformin thrice times daily and low calorie diet for 12 weeks. Group I, additionally will perform one hour of treadmill walking thrice weekly for 12 weeks.
  Interventions: Behavioral: exercise and limiting diet
- group number 2 (Active Comparator): Twenty females with PCOS, eye dryness , and obesity will receive metformin thrice times daily and low calorie diet for 12 weeks.
  Interventions: Behavioral: diet limitation

INTERVENTIONS:
Behavioral: exercise and limiting diet — twenty females with PCOS, eye dryness , and obesity will receive metformin thrice times daily and low calorie diet for 12 weeks. Group I, additionally will perform one hour of treadmill walking thrice weekly for 12 weeks.
  Arms: group number 1
Behavioral: diet limitation — twenty females with PCOS, eye dryness , and obesity will receive metformin thrice times daily and low calorie diet for 12 weeks.
  Arms: group number 2

SUMMARY:
Women with polycystic ovarian syndrome (PCOS) may complain dryness of their eyes especially obese ones. lifestye changes are main treatrment fro both problems

DETAILED DESCRIPTION:
Forty females with PCOS, eye dryness , and obesity will asigned to group I or Group II, n=20 for each group. Both groups will receive metformin thrice times daily and low calorie diet for 12 weeks. Group I, additionally will perform one hour of treadmill walking thrice weekly for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women
* obese class I
* bilateral dryness of eye

Exclusion Criteria:

* liver disoease
* cardiac disease
* renal disease

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
schrimer test | it will be measured after 12 weeks
  it is a test for assessment dye dryness

SECONDARY OUTCOMES:
Ocular surface disability index | It will be measured after 12 weeks
  it is a questionaire for assessment dye dryness
dry eye scoring system | It will be measured after 12 weeks
  it is a questionaire for assessment dye dryness
Tear film break-up time | It will be measured after 12 weeks
  it is a test for assessment dye dryness
body mass index | it will be measured after 12 weeks
  it will be assessed on empty stomach and bowel
wasit hip ratio | It will be measured after 12 weeks
  it will be assessed by dividing wasit circuference on hip circumference
wasit circumference | It will be measured after 12 weeks
  it will be assessed by tape measure
testesterone | It will be measured after 12 weeks
  it will be assessed in serum
LH:FSH ratio | It will be measured after 12 weeks
  The LH (Luteinizing Hormone) to FSH (Follicle-Stimulating Hormone) ratio shows the balance between these reproductive hormones
dehydroepiandrosterone | It will be measured after 12 weeks
  it will ne assessed in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt